CLINICAL TRIAL: NCT06736392
Title: Efficacy of Dexmedetomidine As an Adjuvant to Bupivacaine in Ultrasound Guided Pericapsular Nerve Group Block for Postoperative Analgesia During Spinal Anesthesia in Hip Replacement Surgeries, a Randomized Controlled Study
Brief Title: Efficacy of Dexmedetomidine As an Adjuvant to Bupivacaine in Pericapsular Nerve Group Block in Hip Replacement Surgeries
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mamdooh Wardany, DOCTOR, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dexmedetomidine in PENG block
Record Dates: First submitted 2024-12-08; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: PENG Block
MeSH Terms: interventions — Dexmedetomidine; Needles

STUDY DESIGN:
Intervention Model Description: A calculated minimum sample of 60 patients candidate for hip replacement surgeries (will have spinal anesthesia with hyperbaric bupivacaine 0.5%) will be randomly assigned into one of two equal groups (1:1 design) (Group-C (control) (n=30); will have PENG block using 20ml of isobaric bupivacaine 0.25% and Group-D (n=30); will have PENG block with 1.5μg/kg dexmedetomidine as an adjuvant to 20ml of isobaric bupivacaine 0.25%, to have 80% power to detect an absolute difference of 0.1 in the mean of the postoperative analgesic consumption in nine repeated measures(at 0,2,4,6,8,10,12,16,24 hours postoperatively), at significance level of 0.05.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- group C (Active Comparator): (Group-C (control) (n=30); will have PENG block using 20ml of isobaric bupivacaine 0.25%
  Interventions: Procedure: Ultrasound guided Pericapsular Nerve Group Block; Drug: Isobaric Bupivacaine 0. 25%; Device: the ultrasound machine with curvilinear transducer (high -frequency probe, 2.5Mhz to 7.5Mhz); Device: a standard echogenic 20-22 gauge 100mm needle
- group D (Active Comparator): Group-D (n=30); will have PENG block with 1.5μg/kg dexmedetomidine as an adjuvant to 20ml of isobaric bupivacaine 0.25%
  Interventions: Procedure: Ultrasound guided Pericapsular Nerve Group Block; Drug: 20 ml isobaric bupivacaine 0.25% and 1.5μg/kg dexmedetomidine; Device: the ultrasound machine with curvilinear transducer (high -frequency probe, 2.5Mhz to 7.5Mhz); Device: a standard echogenic 20-22 gauge 100mm needle

INTERVENTIONS:
Procedure: Ultrasound guided Pericapsular Nerve Group Block — With the patient in the supine position and the leg slightly abducted, a curvilinear transducer (2.5-7.5 MHz) is prepared with sterile conduction gel and covered with a sterile probe cover. The transducer is placed transversely over the anterior superior iliac spine (ASIS), then aligned with the pubic ramus and rotated approximately 45° parallel to the inguinal crease. The probe is slid medially to identify key landmarks: the anterior inferior iliac spine (AIIS), iliopubic eminence (IPE), iliopsoas tendon, femoral artery, and femoral nerve. Sliding the probe distally or tilting caudally exposes the femoral head.
  A 20-22 gauge echogenic needle (100 mm) is inserted in-plane from lateral to medial, targeting the plane between the psoas tendon and the pubic ramus. the anesthetic agent is deposited to lift the psoas tendon while avoiding tendon puncture.
Drug: Isobaric Bupivacaine 0. 25% — group c will receive PENG block with only 20ml isobaric bupivacaine 0.25%
  Arms: group C
Drug: 20 ml isobaric bupivacaine 0.25% and 1.5μg/kg dexmedetomidine — group D will receive PENG block with 20 ml isobaric bupivacaine 0.25% and 1.5μg/kg dexmedetomidine
  Arms: group D
Device: the ultrasound machine with curvilinear transducer (high -frequency probe, 2.5Mhz to 7.5Mhz) — the two groups will receive the PENG block under ultrasound guidance
Device: a standard echogenic 20-22 gauge 100mm needle — the two groups will receive the PENG block using a standard echogenic 20-22 gauge 100mm needle

SUMMARY:
Our aim will be to investigate the efficacy of dexmedetomidine as an adjuvant to bupivacaine in ultrasound guided pericapsular nerve group (PENG) block for postoperative analgesia in hip replacement surgeries.

* Our primary outcome of the study: total amount of postoperative morphine consumption in the first 24h postoperative.
* Our secondary outcome of the study: postoperative analgesia assessed by pain score (by Visual Analog Scale)

DETAILED DESCRIPTION:
Effective postoperative pain management is essential for optimizing recovery and patient outcomes following hip surgeries.

The pericapsular nerve group (PENG) block has gained attention as a regional anesthesia technique that provides targeted analgesia to the hip joint and surrounding structures, reducing opioid consumption and avoiding its side effects as nausea, vomiting, constipation, itching, rash, addiction, urinary retention, respiratory depression especially at higher doses By delivering local anesthetics close to the genicular branches of the femoral nerve, the pericapsular nerve group (PENG) block offers several advantages as part of multimodal analgesia in comparison to other nerve blocks used for hip surgeries, such as the femoral nerve block (FNB) and the lumbar plexus block (LPB) as better pain relief for capsular structures with minimal motor blockade, lower risk of complications and reducing need for opioids making it particularly suitable for orthopedic procedures.

Traditionally, local anesthetics such as bupivacaine have been used in the pericapsular nerve group (PENG) block to achieve effective analgesia. However, despite its long acting properties, their duration of action is typically limited to 6 to 12 hours depending on factors like the concentration, dose and individual patient characteristics and the quality of analgesia may diminish as the anesthetic effect wears off, potentially necessitating additional analgesic interventions or systemic opioids to maintain pain control.

Therefore, there is a growing interest in exploring adjuvants that can enhance the efficacy and duration of pain relief without compromising safety such as Dexmedetomidine, Clonidine, and Dexamethasone.

Dexmedetomidine, a highly selective alpha-2 adrenergic agonist, has emerged as a promising adjuvant in prolonging the duration and improving the quality of peripheral nerve blocks through its potent analgesic and sedative effects, by binding to its receptors, reducing the release of norepinephrine and inhibiting pain transmission , by this mechanism not only enhances sensory blockade but also provides effective postoperative analgesia with minimal motor impairment.

Studies have shown that dexmedetomidine, when added to local anesthetics in various regional anesthesia techniques, including peripheral nerve blocks, significantly prolongs the duration of sensory blockade and improves postoperative pain scores.

Given the potential benefits of dexmedetomidine in enhancing postoperative pain management and reducing opioid requirements, this study aims to evaluate its efficacy as an adjuvant to bupivacaine in the pericapsular nerve group (PENG) block for hip replacement surgeries. By assessing, opioid consumption and pain scores, this research seeks to contribute valuable insights into optimizing analgesic strategies in orthopedic anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 years to 90 years
* Gender : both males and females
* BMI less than 35 kg/m2
* Patients with American society of anesthesiologists (ASA) classification class I , II or III
* Patients scheduled for total or partial hip replacement surgery under spinal anesthesia

Exclusion Criteria:

* Patient declining to give written informed consent
* Patient with infection at the site of injection
* Patient with coagulopathy
* Patients with known allergy to used medications.
* Psychiatric disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
total amount of postoperative morphine consumption in the first 24h postoperative. | within the first 24 hours postoperatively

SECONDARY OUTCOMES:
the intensity of postoperative pain assessed by the Visual Analog Scale for pain | within the first 24 hours postoperatively
  the intensity of postoperative pain assessed by the Visual Analog Scale for pain , which was scored from 0 to 10 where 0= no pain and 10 = the worst pain imaginable at 0,2,4,6,8,10,12,16,24 hours post-operatively to evaluate acute pain

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mohamed Abd Ellatif, Study Director — Anesthesia, Intensive Care and Pain management ,Faculty of medicine, Assiut University; Shereen Mamdooh Mohamed, Study Director — Anesthesia, Intensive Care and Pain management South Egypt Cancer Institute, Assiut University; Moaaz Mohamed Tohamy, Study Director — Anesthesia, Intensive Care and Pain management South Egypt Cancer Institute, Assiut University